CLINICAL TRIAL: NCT04466410
Title: A Double Blind, Placebo Controlled, Preliminary Evaluation of Safety, Tolerability, and Efficacy of XT-150 for the Treatment of Neuropathic Pain
Brief Title: Safety and Efficacy of XT-150 for Treatment of Neuropathic Pain
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Failure to enroll a sufficient number of patients.
Sponsor: Xalud Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XT-150-1-0102
Record Dates: First submitted 2020-06-24; First posted 2020-07-10 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Neuropathic Pain
Keywords: XT-150; Plasmid Gene Therapy; IL-10
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Intervention Model Description: Dose escalation by cohort following safety reviews
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo and active drug are identical in appearance. Randomization will be provided to an unblinded pharmacist. Dosing and clinical assessments will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 0.015 milligram (mg) XT-150 (Experimental): 0.015 mg of XT-150. Cohort 1 of the study
  Interventions: Biological: XT-150
- 0.15 mg XT-150 (Experimental): 0.15 mg of XT-150. Cohort 2 of the study
  Interventions: Biological: XT-150
- 0.45 mg XT-150 (Experimental): 0.45 mg of XT-150. Cohort 3 of the study
  Interventions: Biological: XT-150
- Placebo (Placebo Comparator): PBS for injection.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: XT-150 — Single bolus intrathecal injection
  Other Names: IL-10 transgene plasmid DNA injected intrathecally
  Arms: 0.015 milligram (mg) XT-150; 0.15 mg XT-150; 0.45 mg XT-150
Biological: Placebo — Placebo is a sterile phosphate-buffered saline
  Arms: Placebo

SUMMARY:
Preliminary Evaluation of Safety, Tolerability, and Efficacy of XT-150 for the Treatment of Neuropathic Pain. Intrathecally administered, single injection.

DETAILED DESCRIPTION:
XT-150 has been safe and well tolerated in clinical studies of intra-articular knee injections for osteoarthritis.

This is the initial study of XT-150 for treatment of neuropathic pain. For this indication XT-150 must be administered by intrathecal injection. Doses used in the osteoarthritis studies will be studied for neuropathic pain.

Upon safety reviews, doses will be increased by cohorts.

The study is placebo controlled and blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Male or female, between 18 and 80 years of age, inclusive
3. Clinical indication: Lumbar disk disease with no prior lumbar surgery with radicular pain symptoms and/or signs of compressive neuropathy
4. At screening and baseline, a pain intensity score > 60 using the visual analog scale of pain intensity [VASPI] (0-100 mm scale) and a participant reported history of pain in the past 3 or more months
5. Medically stable as determined by the Principal Investigator in consultation with the Sponsor's Medical Monitor, based on pre-study medical history, physical examination, and clinical laboratory tests
6. In the judgment of the Principal Investigator, acceptable vital signs: blood pressure; resting heart rate; respirations, and oral temperature
7. Life expectancy >6 months as determined by the Principal Investigator
8. Female participants of child-bearing potential, and those <1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full menstruation cycle before study drug administration and agree to continue abstinence for 1 full menstruation cycle after the study is completed
9. Male participants who are heterosexually active, and not surgically sterile, must agree to use effective contraception for the duration of the study and for 1 month after the study is completed
10. Stable medical regimen for ≥1 month before screening assessments
11. Have suitable lumbar anatomy for intrathecal injection as determined by MRI or X-Ray in the last 6 months.
12. Willing and able to return for the follow-up (FU) visits
13. Able to read and understand study instructions, and willing and able to comply with all study procedures
14. Adequately informed of the nature and risks of the study and give written informed consent before receiving any study specific assessments or procedures
15. Stable use of non-prescription pain therapy, including massage, TENS, physiotherapy osteopathy, chiropractic and acupuncture for 2 months prior and throughout the study period

Exclusion Criteria:

Participants must NOT meet any of the following exclusion criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of the study drug
2. Any spinal deformity preventing intrathecal injection or making intrathecal injection unsafe
3. Prior history of lumbar surgery, including fusion and microdiscectomy
4. History of epidural block or facet block or steroid injection in the last 6 months
5. Current unstable angina, uncontrolled congestive heart failure, or >1+ pitting edema of lower extremities
6. History of acute myocardial infarction, transient ischemic attack, stroke, or seizure within 3 months of screening visit
7. Severe chronic obstructive or restrictive pulmonary disease
8. Current insulin dependent diabetes mellitus
9. Current autoimmune conditions or documented immunodeficiency
10. History of immunosuppressive therapy; high-potency systemic steroids in the last 3 months
11. Current treatment with systemic immunosuppressive (systemic corticosteroid therapy [equivalent to >10mg/day prednisone] or other strong immunosuppressant)
12. Current or history of central nervous system cancer
13. Any malignancy (EXCEPTION: localized non-melanoma skin cancers) within 5 years before the screening visit or currently receiving systemic chemotherapy, radiation therapy, or a surgical stabilization procedure
14. Significant hepatic disease as indicated by clinical laboratory results for the following: ≥3 times the upper limit of normal (ULN) for aspartate aminotransferase, alanine aminotransferase, ≥ 2.5 time ULN alkaline phosphatase, or ≥1.5 times ULN for total bilirubin)
15. Severe anemia (Grade 3; hemoglobin <8.0 g/dL, <4.9 mmol/L, <80 g/L; transfusion indicated), Grade 1 white cell counts (lymphocytes <LLN - 800/mm3; <LLN - 0.8 x 109 /L, neutrophils <LLN - 1500/mm3; <LLN - 1.5 x 109 /L)
16. Significant renal disease as indicated by creatinine ≥1.5 times the upper limit of normal or creatinine clearance <80 mL/minute (Cockcroft-Gault formula estimate)
17. Confirmed positive for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus
18. Significant psychological conditions; dementia, major depression, or altered mental state that in the opinion of the Investigator will interfere with study participation
19. Current treatment with systemic antibiotics or antivirals (EXCEPTION: topical treatments)
20. Current treatment with anticoagulants /antiplatelet medications except for low dose aspirin or low dose aspirin-containing compounds. Participants, if medically feasible, can interrupt anticoagulant therapy by following local medical practice protocol for intrathecal injections for participants on anticoagulant, antiplatelet therapy.
21. Current use of systemic corticosteroids (equivalent to >10mg/day prednisone)
22. Known or suspected history of active alcohol or illicit drug abuse within 1 year before the screening visit
23. Women who are pregnant or nursing
24. Use of any investigational drug or device within 1 month before randomization or current participation in a trial that included intervention with a drug or device; or currently participating in an investigational drug or device study
25. Any condition that, in the opinion of the Principal Investigator, could compromise the safety of the participants, the participant's ability to communicate the study staff, or the quality of the data
26. Presence of an implanted intrathecal infusion system or peripheral neurostimulator
27. Presence of a generalized pain disorder such as fibromyalgia or complex regional pain syndrome that in the opinion of the PI may impact on evaluation of response to the study drug
28. Diagnosis of peripheral neuropathy of the lower extremities which in the opinion of the PI, might interfere with the participant's ability to assess the effect of the study drug on the radicular signs and/or symptoms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events and Serious Adverse Events | 6 months
Number of participants with abnormal vital signs | 6 months
Number of participants with clinically significant abnormal physical examination findings | 6 months
Number of participants with anti-interleukin (IL)-10 antibodies | 6 months
Number of participants with IL-10 Protein | 6 months
Number of participants with abnormal clinical and hematology parameters | 6 months
Number of participants with plasmid DNA present in whole blood | 6 months
Number of participants with cytokines in Cerebrospinal fluid | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Howard Rutman, MD,MBA, Study Director — Xalud Therapeutics, Inc.
Locations (4):
- Australia (4):
  - Genesis Research Services, Newcastle, New South Wales
  - CerCare, Wayville, South Australia
  - Metro Pain Group, Clayton, Victoria
  - Alfred Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No